CLINICAL TRIAL: NCT05382897
Title: Effects of a Fasting Mimicking Diet on Depressive Symptoms in Patients With Inflammatory Bowel Disease
Brief Title: Fasting-mimicking Diet in Treatment of Depressive Symptoms in IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: W. Garfield Weston Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00115405
Record Dates: First submitted 2022-01-31; First posted 2022-05-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: depression; diet; microbiome; fasting; inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Depression; Fasting

STUDY DESIGN:
Intervention Model Description: This is an exploratory randomized double-blind parallel trial using a fasting-mimicking diet (FMD) in patients with inflammatory bowel disease (IBD) who are in clinical remission but experiencing depression
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator and lab personnel involved in assessment of outcomes will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting-Mimicking Diet (Experimental): Participants will be followed for 3 weeks for baseline assessment and then consume a plant-based fasting-mimicking diet for 5 days once a month for 3 months.
  Interventions: Other: Plant-based fasting-mimicking diet
- Caloric-Sufficient Diet (Experimental): Participants will be followed for 3 weeks for baseline assessment and then consume a plant-based caloric-sufficient diet for 5 days once a month for 3 months.
  Interventions: Other: Plant-based fasting-mimicking diet

INTERVENTIONS:
Other: Plant-based fasting-mimicking diet — Participants will be on a low caloric plant-based diet or a caloric-sufficient plant-based diet for 3 x 5 day cycle each month followed by 3 weeks of eating normally for a total period of 3 months.

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic illness characterized by inflammation of the intestine. Many individuals with IBD suffer from depressive symptoms and anxiety which can lead to a decreased quality of life, poor treatment compliance, and higher morbidity and mortality. The object of this clinical trial is to investigate the effects of a fasting mimicking diet in IBD patients who are suffering with symptoms of depression. Participants will carry out 3 cycles of a 5-day period of a plant-based low caloric diet or a plant-based caloric sufficient diet following by 3 weeks of eating normally. Effects of the dietary intervention on microbes in the gut, immune and metabolic function, and depressive symptoms will be measured. The overall goal is to develop a safe and effective treatment to improve mental health in patients with IBD by targeting the gut microbiome through dietary interventions.

DETAILED DESCRIPTION:
The primary objective of this proof of principle study is to investigate the effects of a fasting mimicking diet on depressive symptoms in patients with inflammatory bowel disease.

The specific aims of this project include:

1. Determine whether a fasting-mimicking diet is effective in ameliorating depressive symptoms in patients with Crohn's disease or ulcerative colitis
2. Determine if beneficial effects seen during the interventional period are sustained following cessation of fasting
3. Examine effects of the intervention on the gut microbiome and metabolome

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 65 years at the time of screening
* Diagnosis of Crohn's disease in clinical remission or with mild-moderate disease with Harvey Bradshaw Index (HBI<8) or diagnosis of ulcerative colitis in clinical remission with partial Mayo (pMayo<7)
* Suffering from mild-moderate depression with PHQ-9 ≥5 and ≤ 19

Exclusion Criteria:

* Subjects who are reliant on partial or total parenteral nutrition
* Subjects with prior gastrointestinal surgery and consequences such as short bowel syndrome, ostomy of small or large intestine, total colectomy, proctocolectomy, or ileoanal pouch
* Subjects with diabetes or celiac disease
* Subjects with a body mass index (BMI) lower than 18
* Subjects suffering from malnutrition or at high risk of malnutrition assessed by a score of ≥6 on the abridged patient generated subjective global assessment (PGSGA)
* Subjects allergic to nuts
* Subjects currently on a fasting/intermittent type caloric restricted diet
* History of psychotic or bipolar disorders or experiencing suicidal thoughts
* Pregnant women, women who are breast feeding, or women planning on becoming pregnant
* Subjects with immune-compromised condition other than inflammatory bowel disease (e.g. AIDS, lymphoma)
* Subjects with severe uncontrolled cardiovascular or respiratory disease or active malignancy
* Unable to read English or provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Changes in Patient Health Questionnaire (PHQ-9) | From baseline through 12 and 24 weeks
  A change in depressive symptoms as assessed through the Patient Health Questionnaire (PHQ)-9. [Min:0; Max 27; good to poor]

SECONDARY OUTCOMES:
Changes in Harvey-Bradshaw Index (HBI) in patients with Crohn's disease | From baseline through 12 and 24 weeks
  Changes in disease status as assessed by HBI in Crohn's disease patients
Changes in partial Mayo Score in patients with ulcerative colitis | From baseline through 12 and 24 weeks
  Changes in disease status as assessed by partial Mayo Score in patients with ulcerative colitis
Changes in clinical markers of disease | From baseline through 12 and 24 weeks
  Changes in serum C-reactive protein (CRP)
Changes in clinical markers of disease | From baseline through 12 and 24 weeks
  Changes in fecal calprotectin
Changes in levels of fatigue | From baseline through 12 and 24 weeks
  Changes in level of fatigue as assessed by the inflammatory bowel disease-fatigue (IBD-F) self-assessment scale (0-20; low to high)
Changes in general anxiety | From baseline through 12 and 24 weeks
  Changes in general anxiety as assessed by the Hospital Anxiety and Depression scale (HADS) (0-21; low to high)
Changes in quality of Life | From baseline through 12 and 24 weeks
  Changes in quality of life as assessed by Short Inflammatory Bowel Disease Questionnaire (SIBDQ) (score 10-70, poor to good)
Changes in weight | From baseline through 12 and 24 weeks
  Changes in weight in kilograms
Changes in body mass index (BMI) | From baseline through 12 and 24 weeks
  Changes in BMI as assessed by weight in kilograms divided by the square of height in meters
Changes in gene expression in peripheral blood mononuclear cells | From baseline through 12 and 24 weeks
  Changes in immune function as assessed by changes in gene expression of peripheral blood mononuclear cells
Changes in blood cytokines | From baseline through 12 and 24 weeks
  Changes in plasma concentrations of cytokines (TNF, IL-6, IL-8, IFNγ, IL-1β, IL-9, IL-10, IL-12, IL-17, TGFβ)
Changes in blood hormones | From baseline through 12 and 24 weeks
  Changes in plasma concentrations of hormones (ghrelin, leptin, BDNF, GLP-1, glucagon, insulin)
Changes in gut microbiome | From baseline through 12 and 24 weeks
  Changes in gut microbiome as assessed by 16s rRNA analysis
Changes in fecal short chain fatty acids | From baseline through 12 and 24 weeks
  Changes in fecal concentrations of short chain fatty acids
Changes in fecal bile acids | From baseline through 12 and 24 weeks
  Changes in fecal concentrations of primary and secondary bile acids

CONTACTS AND LOCATIONS:
Overall Officials: Karen Madsen, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Alberta Human Nutrition Research Unit, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No